CLINICAL TRIAL: NCT00931489
Title: Retinal and RPE Autoimmunity in AMD: Assessment of Correlation With Degree of Response to Ranibizumab Therapy
Brief Title: Retinal and Retinal Pigment Epithelium (RPE) Autoimmunity in Age-related Macular Degeneration (AMD)
Acronym: Antibody
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lawrence S. Morse, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lawrence S. Morse, MD, Professor, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 217330; FVF4479s (Other: Genentech)
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Age Related Macular Degeneration
Keywords: Age Related Macular Degeneration; Lucentis; Ranibizumab; Antibodies; Retinal and RPE Autoimmunity
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Wet AMD Patients Responders (Active Comparator): Dilated eye exam once a month for 7 months; visual acuity and OCT once a month for 7 months; Lucentis(R)/ranibizumab injection once each month for the Baseline and Month 1-3 visits, then as needed at Month 4 and 5; 3 Tbls. blood draw at Baseline, Month 3 and Month 6 visits.
  Interventions: Drug: ranibizumab (Lucentis(R))
- Normal Population (No Intervention): Dilated eye exam and 3 Tbls. blood draw at first and only study visit.
- Wet AMD Patients Acute Non-responders (Active Comparator): Participants in this Group will have not responded to 4 prior injections of Lucentis(R)/ranibizumab or other anti-VEGF treatment. Dilated eye exam at Month 4; visual acuity and OCT at Months 4-6; injection of anti-VEGF treatment as needed at Months 4 and 5; 3 Tbls. blood draw at Month 4
  Interventions: Drug: ranibizumab (Lucentis(R))
- Dry AMD Population (No Intervention): Dilated eye exam and 3 Tbls. blood draw at first and only study visit.
- Wet AMD Patients Chronic Non-responderes (Active Comparator): Participants in this Group will have not responded to 4 or more prior injections of Lucentis(R)/ranibizumab or other anti-VEGF treatment. One visit at Month 4: Dilated eye exam with visual acuity and OCT; injection of anti-VEGF as needed; 3 Tbls. blood drawn
  Interventions: Drug: ranibizumab (Lucentis(R))

INTERVENTIONS:
Drug: ranibizumab (Lucentis(R)) — 0.5 mg intravitreal injection once a month for 4 months, then as needed for 2 months
  Other Names: Lucentis(R)
  Arms: Wet AMD Patients Acute Non-responders; Wet AMD Patients Chronic Non-responderes; Wet AMD Patients Responders

SUMMARY:
The investigators hope to determine if "wet" AMD patients differ from patients with "dry" AMD or normal eyes in the production of anti-retinal pigment epithelium (anti-RPE) or anti-retinal antibody formation. To explain: the immune system can make antibodies that attack our own cells, specifically the RPE and the retina. Normally the RPE and retinal cells are ignored by the immune system, but when disease occurs, immune reactions can occur, making an autoantibody that can attack the patient's own cells and make things worse. This production of autoantibodies that react with our own RPE and retinal cells is what the investigators want to test in this proposal to see if they may contribute to, or are responsible for, a poor response to treatment.

The investigators also want to know how those patients who initially respond to the standard-of-care treatment, ranibizumab injections, differ in the production of anti-RPE or anti-retinal antibody formation, from those patients who do not respond initially after 4 consecutive injections.

DETAILED DESCRIPTION:
Up to 10% of patients with neovascular AMD treated with ranibizumab respond poorly or worsen despite therapy. The reason for this lack of response is unclear. We have preliminary data that suggests abnormal autoimmune activity is apparent in these patients. Previous studies have shown evidence of retinal autoimmunity in AMD patients, but there is very little data describing any specific immunologic commonality that correlates with disease and/or poor response. (8,9) Perhaps just as significantly there is little data regarding the immunologic activity of age-matched normals, making published data hard to evaluate especially in this age group in which autoimmunity is known to increase. (8,9) While there are many known retinal antigens in autoimmune retinal disease, the role of these antigens is not well established in AMD and not all the antigens have been identified. (24) Moreover, RPE-reactivities are only beginning to be understood in ocular disease. (25-27) We intend to address humoral responses in AMD by making a systematic comparison of the immunologic activity of ranibizumab responders, ranibizumab initial non-responders, and a comparable population of age-sex-race matched normal controls. Data suggests that 5 groups of patients are evident after 3 treatments with ranibizumab: 1) rapid responders, 2) delayed responders, 3) gradual responders, 4) acutenon-responders and 5) chronic non-responders. We hypothesize that non-responders and gradual responders may in fact be patients with complicating underlying autoimmune activity involving retinal and RPE antigens, which are exposed secondary to the breakdown of the blood-retinal barrier during CNV development. We will study this humoral response (antibody production) over the treatment period, as it likely is changing at different rates in the patients with different responses. In addition we will correlate underlying genetic phenotype in these patients.

For this study, we plan to look at 2 treatment groups and 2 control groups:

* Group 1: patients with neovascular AMD who respond to ranibizumab after 4 consecutive injections with ranibizumab
* Group 2: age-sex-race matched normal population controls (without AMD)
* Group 3: patients with neovascular AMD who are acute non-responders to anti-VEGF treatment after 4 or more consecutive injections
* Group 4: age-sex-race matched dry AMD patients (AREDS category 2/3 ou) controls
* Group 5: patients with neovascular AMD who are chronic non-responders to anti-VEGF treatment after 4 or more consecutive injections

This is an open-label study assessing antibody formation (anti-RPE and anti-retinal) in 5 groups. Group 1 (n=40) will include neovascular AMD patients treated with ranibizumab. Patients will be included and receive 4 ranibizumab 0.5mg intravitreally at 4-6 week intervals and then twice more "as needed" (PRN) at 4-6 week intervals. After the 4th ranibizumab injection, if a Group 1 patient has not responded (persistent fluid on OCT), they will be moved into Group 3 (anti-VEGF acute non-responders) or Group 5 (anti-VEGF chronic non-responders). This will reduce the eventual number of subjects enrolled in Group 1 to approximately 36, as we anticipate approximately 4 subjects to have to move to either Group 3 or Group 5 as a non-responder. Group 2 (n=40) will be an age-sex-race matched normal subjects from the population that does not have AMD. Group 3 (n=8) and Group 5 (n=7) (for a combined total of 15 subjects, approximately 4 of whom transferred from Group 1) include patients treated with 4 or more injections of anti-VEGF treatment at 4-8 week intervals without an initial response (Initial non-response is defined as < 100 microns of improved [decreased] retinal thickening by OCT). Group 3 patients, the acute non-responders, will be included after the 4th injection and followed for 2 more visits at 4-8 week intervals during which time they can receive "as needed" anti-VEGF treatment(s) at the investigator's discretion for any fluid on OCT. Group 4 (n=40) will be age-sex-race matched patients with Dry AMD as controls for immune response before there is a neovascular response. Group 5 patients, the chronic non-responders, will be included after the 4th injection and followed for one (1) visit at Month 4 during which time they can receive an "as needed" anti-VEGF treatment at the investigator's discretion for any fluid on OCT.

NOTE: Only 10% of Group 1 (approximately 4 patients) are expected to be non-responders, therefore, 11 of the Group 3 and Group 5 subjects will be patients treated outside the study who are found to be non-responders by chart review. These patients will then be enrolled at the Month 4 visit to supplement the subjects transferred from Group 1 for a total of 15 patients in Groups 3 and 5.

We will use Western blotting for global assessment of all autoantibodies against the full complement of retinal proteins in both normal individuals (Group 2) and those treated for exudative AMD (Group 1), those initial non-responders to ranibizumab (Group 3), and patients with "dry" AMD (Group 4).

Genotyping (CFH and HTRA1) will be performed on all Groups. Approximately 25 ml (2 tablespoons) of blood will be sent to Dr. Khang Zhang of the Shiley Eye Center at the University of California, San Diego and he will perform the genetics analysis.

This study will investigate if antibody production differs between nv AMD patients (Groups 1, 3 and 5) and the normal population (Group 2), if it differs between ranibizumab responders (Group 1) and non-responders to any anti-VEGF treatment (Groups 3 and 5), and we will also see how patients with dry AMD (Group 4) compare with the nv AMD groups (Groups 1, 3, and 5).

ELIGIBILITY:
Inclusion Criteria:

* Group 1 (Ranibizumab Responders):

  * Ability to provide written informed consent and comply with study assessments for the full duration of the study
  * Age > 50 years
  * Patients with active neovascular "wet" AMD naïve to treatment
* Group 2 (Normal Controls):

  * Age-sex-race matched to Group 1 patients
  * Non-AMD
  * Ability to provide written informed consent
* Group 3 (Anti-VEGF Initial Non-responders):

  * "Wet" AMD patient treated with 4 or more monthly injections of anti-VEGF treatment without an adequate response (persistent fluid on OCT)
  * Ability to provide written informed consent and comply with study assessments for the full duration of the study
  * Age > 50 years
* Group 4 ("Dry" AMD):

  * Age-sex-race matched to Group 1 patients
  * "Dry" AMD, category 2 or 3 by AREDS (Age-Related Eye Disease Study) criteria
  * Ability to provide written informed consent

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* Concurrent eye disease in the study eye that could compromise visual acuity (e.g., diabetic retinopathy, advanced glaucoma)
* Previous AMD therapy
* Patients being treated for autoimmune or other disease with immunomodulatory drugs (i.e., prednisone, infliximab, methotrexate)
* Patients with recent (less than 6 months) ocular or systemic surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2009-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence S Morse, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Wet AMD Patients Chronic Non-responderes: Participants in this Group will have not responded to 4 or more prior injections of anti-VEGF treatment. One visit at Month 4: Dilated eye exam with visual acuity and OCT; injection of anti-VEGF as needed; 3 Tbls. blood drawn
  ranibizumab (Lucentis(R)): 0.5 mg intravitreal injection once a month for 4 months, then as needed for 2 months
Period: Overall Study
Arm/Group | Wet AMD Patients Responders | Normal Population | Wet AMD Patients Acute Non-responders | Dry AMD Population | Wet AMD Patients Chronic Non-responderes
Started | 40 | 40 | 5 | 39 | 7
Completed | 40 | 40 | 5 (3 subjects enrolled in Group 1 (responders) were moved to Group 3 (non-responders)) | 39 | 7
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Acute Non-responders (Group 3) had 5 subjects at baseline but increased at 6 month timepoint because 3 subjects originally enrolled into Group 1 (Responders) were deemed "non-responders" (had persistent subretinal fluid on Ocular Coherence Tomography) and were moved to Group 3.
Groups:
- Total: Total of all reporting groups
Arm/Group | Wet AMD Patients Responders | Normal Population | Wet AMD Patients Acute Non-responders | Dry AMD Population | Wet AMD Patients Chronic Non-responderes | Total
Number analyzed (Participants) | 40 | 40 | 5 | 39 | 7 | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 80.35 (9.24) | 67.82 (7.39) | 78.20 (8.41) | 77.08 (9.50) | 82.86 (8.41) | 75.60 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 3 | 22 | 3 | 75
  Male | 16 | 17 | 2 | 17 | 4 | 56

OUTCOME MEASURES:

1. Primary Outcome: Production of Anti-Retinal Pigment Epithelium (RPE) or Anti-retinal Antibody Formation in Neovascular ("Wet") Age-related Macular Degeneration Patients Compared to Population Normals.
Description: Blood samples were collected from all study participants at baseline and Western Blot analysis was performed to identify the presence of anti-retinal and anti-RPE antibodies. Presented are the number of subjects in which the presence of anti-retinal and anti-RPE antibodies (yes/no) were recorded by a masked observer.
Time Frame: 6 months
Population: The "wet" AMD patients' 6 month values in production of RPE or anti-retinal antibody formation are being compared to the Normal Population baseline values.
Measure: Number; unit: participants
Groups:
- Neovascular "Wet" Age-related Macular Degeneration Patients: Subjects with active neovascular ("wet") AMD. This includes the subjects that responded to treatment (Ranibizumab 0.5mg intravitreal injections at four week intervals) Group 1, and chronic "non-responders" - those subjects who received four or more anti-VEGF intravitreal injections with persistent fluid on OCT, Group 3.
  At baseline, 40 subjects were enrolled into Group 1 Following 4 months of treatment, 3 subjects were moved to Group 3.
- Population Normals: Normals are subjects that do not have Age-related Macular Degeneration. Group 2
Arm/Group | Neovascular "Wet" Age-related Macular Degeneration Patients | Population Normals
Number analyzed (Participants) | 45 | 40
participants
  Baseline: number analyzed (Participants) | 45 | 39
  Baseline | 31 | 26
  6 Months: number analyzed (Participants) | 43 | 0
  6 Months | 36 |

2. Secondary Outcome: Change in Visual Acuity (VA) From Baseline to Month 6
Description: Subjects visual acuity (VA) was tested using Early Treatment Diabetic Retinopathy Study (ETDRS) charts. Letters correctly read on ETDRS chart was recorded at baseline and 6 months. Mean change was measured.
Time Frame: 6 months
Population: At the 6 month timepoint - 3 of the 40 subjects enrolled into Group 1 (Wet AMD responders) had been moved to Group 3 due to persistent subretinal fluid on OCT (protocol definition of "non-responder" following 4 months of treatment).
Measure: Mean (Full Range); unit: letters gained
Groups:
- Neovascular "Wet" AMD Patients - Responders: Subjects with neovascular ("wet") Age-related Macular Degeneration who respond to ranibizumab after 4 consecutive intraocular injections Group 1
- Neovascular "Wet" AMD Patients - Acute Non-responders: Subjects with neovascular ("wet") AMD treated with 4 or more monthly injections of anti-VEGF without an adequate response (persistent fluid on OCT) Group 3 - non-responders
Arm/Group | Neovascular "Wet" AMD Patients - Responders | Neovascular "Wet" AMD Patients - Acute Non-responders
Number analyzed (Participants) | 37 | 8
letters gained | 10.08 [-10 to 44] | 6.14 [1 to 12]

3. Secondary Outcome: Change in Ocular Coherence Tomography (OCT) From Baseline to Month 6
Description: Ocular Coherence Tomography (OCT) was used to measure retinal central foveal thickness. The mean change from baseline to 6 months was determined and recorded in micrometers (µm).
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Full Range); unit: µm
Arm/Group | Neovascular "Wet" AMD Patients - Responders | Neovascular "Wet" AMD Patients - Acute Non-responders
Number analyzed (Participants) | 37 | 8
µm | -82 [-472 to 35] | 22 [-72 to 171]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Wet AMD Patients Responders | Normal Population | Wet AMD Patients Acute Non-responders | Dry AMD Population | Wet AMD Patients Chronic Non-responderes
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/40 | 0/5 | 0/40 | 0/7
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/5 | 0/40 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wet AMD Patients Responders (N=40) | Normal Population (N=40) | Wet AMD Patients Acute Non-responders (N=5) | Dry AMD Population (N=40) | Wet AMD Patients Chronic Non-responderes (N=7)
Uveitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Uveitis/presumed endophthalmitis, left eye (non-study eye)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No